CLINICAL TRIAL: NCT04797286
Title: Sildenafil for Early Pulmonary Vascular Disease in Scleroderma
Acronym: SEPVADIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00265164
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Scleroderma; Mildly Elevated Pulmonary Pressures
Keywords: SSc-MEP
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Experimental): Sildenafil 20 mg by mouth three(3) times each day
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo by mouth three(3) times each day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 20 mg three times a day. This is the approved dose for the treatment of pulmonary arterial hypertension. It is being studied in this trial with a population who has mildly elevated pulmonary pressures.
  Other Names: Revatio, Viagra
  Arms: Sildenafil
Other: Placebo — Oral pill placebo.
  Arms: Placebo

SUMMARY:
This is a Phase II randomized, double-blind, placebo-controlled trial of sildenafil in men and women with Scleroderma with mildly elevated pulmonary pressures (SSc-MEP) to determine whether sildenafil may be an effective treatment for SSc-MEP.

DETAILED DESCRIPTION:
Data shows that sildenafil (SIL) is an effective therapy in SSc-PAH. SIL has been safely used in many patients with various vascular and cardiovascular diseases over the past three decades. Randomized controlled trial data for SIL shows improvement in 6MWD, hemodynamics, and even evidence of cardiac remodeling in PAH and SSc-PAH patients. Based upon these data, SIL may be an effective therapy in SSc-MEP. This study will help determine whether sildenafil could be a good treatment for patients with scleroderma that have mildly elevated pulmonary pressures.

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure between 21 and 24 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) ≤ 15 mm Hg within six months before study entry.
* Diagnosis of SSc according to 2013 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) classification criteria.
* Pulmonary function tests with forced expiratory volume in one second/forced vital capacity (FEV1/FVC) >50% AND either a) total lung capacity (TLC) or forced vital capacity (FVC) > 70% predicted or b) TLC or FVC between 60% and 70% predicted with no more than mild interstitial lung disease on computerized tomography scan of the chest on studies obtained within 6 months of enrollment.
* Ventilation perfusion scan or computed tomography with intravenous contrast (CT angiogram) without evidence of chronic thromboembolism at anytime before study entry.
* Ability to perform six minute walk testing without significant limitations in musculoskeletal function or coordination.
* Informed consent.

Exclusion Criteria:

* World Health Organization (WHO) Class IV functional status.
* Systolic blood pressure less than 90 mmHg at screening visit prior to enrollment.
* Clinically significant untreated sleep apnea.
* Left-sided valvular disease (more than moderate mitral valve stenosis or insufficiency or aortic stenosis or insufficiency), pulmonary artery or valve stenosis, or ejection fraction < 45% on most recent echocardiography (within 1 year).
* Use of Pulmonary Arterial Hypertension (PAH) therapy (prostacyclin analogues, endothelin-1 receptor antagonists,phosphodiesterase-5 inhibitors, riociguat, selexipag) within the past 3 months.
* Hospitalized or acutely ill.
* Renal failure (creatinine above 2.0) at screening visit.
* Enrollment in a clinical trial or concurrent use of another investigational drug (non FDA approved) or device therapy within 30 days of screening visit.
* Age < 18.
* Currently pregnant.
* Current use of nitrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change in distance walked in 6 minute walk test (6MWT) at 4 months | Baseline and 4 months
  As assessed by change in 6 minute walk distance (6MWD) in feet (from baseline to 4 months) between the sildenafil group and the placebo group.

SECONDARY OUTCOMES:
Difference in change in distance walked in 6MWT at 12 months | Baseline and 12 months
  As assessed by change in 6 minute walk test distance in feet (from baseline to 12 months) between the sildenafil group and the placebo group.
Difference in change in right ventricular function as assessed by cardiac MRI | Baseline and 4 months
  As assessed by change in right ventricular function (normal/abnormal) on cardiac MRI.
Difference in change in right ventricular function as assessed by cardiac MRI | Baseline and 12 months
  As assessed by change in right ventricular function (normal/abnormal) on cardiac MRI.
Difference in change in right ventricular function as assessed by invasive hemodynamics | Baseline and 4 months
  As assessed by change in right ventricular function (normal/abnormal) on invasive hemodynamics.
Difference in change in right ventricular function as assessed by invasive hemodynamics | Baseline and 12 months
  As assessed by change in right ventricular function (normal/abnormal) on invasive hemodynamics.
Difference in change in right ventricular function as assessed by echocardiography | Baseline and 4 months
  As assessed by change in right ventricular function (normal/abnormal) on echocardiography.
Difference in change in right ventricular function as assessed by echocardiography | Baseline and 12 months
  As assessed by change in right ventricular function (normal/abnormal) on echocardiography.
Difference in change in N-terminal pro b-type natriuretic peptide level | Baseline, 4 months and 12 months
  As assessed by changes in plasma N-terminal pro b-type natriuretic peptide (NT-proBNP) level (pg/mL) between sildenafil and placebo groups at four months and twelve months.
Difference in change in health related quality of life as assessed by the 36-Item Short Form Health Survey (SF36) questionnaire | Baseline, 4 months and 12 months
  As assessed by changes in SF36 questionnaire between sildenafil and placebo groups at four months and twelve months. The SF36 yields a set of scaled scores in 8 domains, with higher numbers representing a better quality of life. Each scale is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Difference in change in health related quality of life as assessed by the emPHasis-10 health-related quality of life questionnaire (emPHasis-10). | Baseline, 4 months and 12 months
  As assessed by changes in emPHasis-10 questionnaire between sildenafil and placebo groups. The Emphasis 10 score consists of 10 questions scored in a semantic 6-point scale (from 0 to 5), for a total maximum score of 50 (the higher the score, the worse the quality of life).
Difference in safety profile as assessed by frequency of adverse events | Ongoing until study closes, up to 4 years
  As assessed by frequency of adverse events between sildenafil and placebo groups.
Difference in safety profile as assessed by severity of adverse events | Ongoing until study closes, up to 4 years
  As assessed by severity of adverse events between sildenafil and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Mathai, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Louisiana State University, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lammi MR, Mukherjee M, Saketkoo LA, Carey K, Hummers L, Hsu S, Krishnan A, Sandi M, Shah AA, Zimmerman SL, Hassoun PM, Mathai SC. Sildenafil Versus Placebo for Early Pulmonary Vascular Disease in Scleroderma (SEPVADIS): protocol for a randomized controlled trial. BMC Pulm Med. 2024 Apr 30;24(1):211. doi: 10.1186/s12890-024-02892-3. PMID 38689245